**Title**: Short versus Long antibiotic course for pleural Infection Management (SLIM trial): protocol of a randomized controlled open label trial

**Version and date:** Version 1.3 – 13<sup>th</sup> Oct 2020

# **Sponsor:**

Alexandria University Faculty of Medicine and Alexandria University Hospitals

Champlion Street, Azarita, Alexandria, Egypt

# Study personnel:

Principal investigator

Dr Maged Hassan

**Lecturer of Chest Diseases** 

Alexandria University Faculty of Medicine

Study co-investigator

Dr Ahmed S Sadaka

**Lecturer of Chest Diseases** 

Alexandria University Faculty of Medicine

**Ethics approval:** the protocol of the study was approved by the Alexandria University Faculty of Medicine Ethics Committee (ref 0304785)

**Registration:** pending (protocol to be submitted to an open-access registry)

### Introduction

Infection of the pleural space is serious condition that requires hospitalization, invasive interventions and long courses of antibiotics<sup>[1]</sup>. Treatment of pleural infection requires long hospital admission with a median of 19 days<sup>[2]</sup> and medical treatments fails requiring surgical intervention in up to 30% of cases<sup>[3]</sup>. The mortality from pleural infection is around 10% at 3 months<sup>[4]</sup>.

Besides drainage of the infected fluid, antibiotics are a core component of management of pleural infection<sup>[5]</sup> and are typically given intravenously in the first few days of treatment until the condition is stabilized at which stage patients are shifted to oral antibiotics of equivalent spectrum. In almost half of the cases of pleural infection, the choice of antibiotics is entirely empirical due to low yield of microbiological tests on pleural fluid in these cases<sup>[6]</sup>. International guidelines cite a minimum length of antibiotic course of pleural infection of four weeks<sup>[5,7]</sup> with antibiotic courses typically lasting six weeks<sup>[8]</sup>. However, these recommendations are based on expert opinion with no robust evidence to support such durations. A recent trial compared a two-week versus a three-week antibiotic course for parapneumonic pleural infections. The trial that concluded prematurely due to inability to recruit to target sample size and found that the two regimens were equivalent in terms of risk of failure of medical treatment<sup>[9]</sup>. Besides being an underpowered study, the results are only applicable to parapneumonic effusions but not primary pleural infections.

The RAPID score has recently been validated as a robust tool to predict 3-month mortality of patients with pleural infection based on demographic and laboratory data (table 1)<sup>[4]</sup>. A low score (0-2) is associated with 2-3% mortality, medium score (3-4) 9% mortality and high score (5-7) 30% mortality at three months<sup>[10]</sup>. The utility for this score in clinical management is yet to be determined and this study will attempt using this score to stratify lengths of antibiotic treatment based on proposed risk of adverse outcomes as stipulated by the RAPID score. A shorter antibiotic course that is as effective as the standard long course is desirable given the common occurrence of side effects with antibiotic treatment. The presence of a robust predictive score of outcome seems as an attractive tool to help stratify patients who can be safely treated with shorter antibiotic courses.

The aim of this study is to investigate the feasibility and safety of prescribing shorter courses of antibiotics (2-3 weeks) versus the standard longer courses (4-6 weeks) in medically-treated patients with pleural infection at lower risk of mortality (RAPID score 0–4) who can be safely discharged home within 14 days of hospitalization and how this impacts success of medical treatment.

Table 1: Components of the RAPID score<sup>[4]</sup>

| Parameter | Value | Score |
|----------------------------|--------------------|-------|
| Renal function | <14 mg/dL | 0 |
| (blood urea nitrogen) | 14-23 mg/dL | 1 |
| | >23 mg/dL | 2 |
| Age | < 50 years | 0 |
| | 50 – 70 years | 1 |
| | > 70 years | 2 |
| Purulence of pleural fluid | Purulent | 0 |
| | Non-purulent | 1 |
| Infection Source | Community-acquired | 0 |
| | Hospital-acquired | 1 |
| Dietary factors | ≥2.7 g/dL | 0 |
| (serum albumin) | <2.7 g/dL | 1 |

#### Methods

This protocol is written in accordance with the guidance of the Standard Protocol Items: Recommendations for Interventional Trials (SPIRIT)<sup>[11]</sup>.

# Trial design and study setting

SLIM is an open label randomized controlled clinical trial that will recruit patients admitted with pleural infection to a University Hospital. Consecutive patients admitted with pleural infection will be invited to take part in an observational study (the Pleural Infection Cohort Study) and consenting to SLIM will occur at the same time of consenting to the cohort study. This design is termed trials within cohorts.<sup>[12]</sup>

Inclusion of other hospitals as recruiting sites is not planned but will be considered if recruitment is deemed slow.

# Eligibility criteria

#### Inclusion

- Adult patients (≥18 years old)
- Willing to provide informed consent
- Admitted to hospital for treatment of pleural infection (both parapneumonic and primary pleural infections included). Pleural infection will be defined by the presence of one of the following:
  - a) the presence of pus in the pleural space;
  - b) positive pleural fluid gram stain or culture; or
  - c) pleural fluid pH < 7.2 or pleural fluid glucose < 40 mg/dL in the setting of acute respiratory infection.
- RAPID low or intermediate score (0-4)
- Fit for discharge within 14<sup>th</sup> day of admission

### Exclusion:

- Failure of medical treatment within 14 days of admission and need for surgical referral
- Need for hospital admission beyond 14 days due to medical reasons
- Admission to recurrent ipsilateral pleural infection within the last three months
- RAPID high score (5 or more)
- Pleural infection not amenable to drainage at time of diagnosis and therefore upfront decision to treat with prolonged antibiotics
- Residual pleural collection (despite attempted drainage) that the managing clinician indicated is for prolonged oral suppressive therapy (i.e. six weeks of oral antibiotics).

Patients will only be randomised to one of the study arms of SLIM if found eligible, and for ineligible patients, their data collection will follow the protocol of the cohort study with no change in their care.

# **Interventions**

The study intervention is the modification of the length of the antibiotic course at the point of discharge from hospital. All other aspects of care will be carried out according to recognised clinical standards. The choice of the antibiotics will rely on results of microbiological studies, and if non-informative will follow international guidelines for treating pleural infection and local patterns of microbiology<sup>[1,6]</sup>. A separate document will be prepared to provide guidance for outpatient antibiotics in the absence of culture results.

In the active arm, patients who are ready for discharge will be prescribed an oral antibiotic course for a minimum period of 7 days and a maximum period that makes the overall length of antibiotic administration 21 days (total number of antibiotic days 14-21 days). In the control arm, at the point of discharge, patients will be prescribed an oral antibiotic course for a minimum of 14 days and a maximum period that makes the overall length of antibiotic administration 42 days (total number of antibiotic days 28-42 days). Treatment duration allocation will be open label.

# Baseline data

Besides patient demographics and infection source, the following data will be collected at the points of admission and discharge as appropriate:

- Date of admission
- Vital signs
- -Blood investigations (minimum: urea and electrolytes, full blood count, C-reactive protein, and serum albumin)
- Pleural fluid parameters (macroscopic appearance, biochemistry, cultures (blood and pleural fluid), pH)
- Chest X-ray at baseline and at discharge
- Thoracic ultrasound (TUS) images at baseline (effusion size and extent of septations)
- Chest computed tomography images at baseline (presence of pleural split sign, lung consolidation or microbubbles)
- Treatments received as inpatient (chest tube size and time till removal, volume of effusion drained, intravenous and oral antibiotics given)
- Total length of hospital admission

# Participant timeline:

Participants admitted to hospital for treatment of pleural infection will be approached to take part in both the observational and interventional studies. For patients who sign an informed consent to both, and upon confirmation of their eligibility to the trial, they will be randomised to a study arm once a decision is made about fitness for discharge from hospital which is within 14 days from admission.

Upon discharge, two face-to-face follow up visits will be planned to coincide with clinical practice of following up patients post admission for pleural infection.

a- Two weeks post discharge (+/- 7 days)

A clinical review to ascertain adherence to treatment and ensure no symptoms of recurrence are present (fever, night sweats, haemoptysis or purulent expectoration, chest pain). Any adverse events related to antibiotic treatment will be recorded. During this visit thoracic US (TUS) +/- chest X-ray will be performed. If a participant is not willing or able to attend in person, a remote review will be performed (via telephone).

b- Six weeks from initial admission (+/- 7 days)

During this visit the following will be performed:

Clinical review of symptoms (relating to infection recurrence or adverse events due to antibiotic treatment)

Check adherence to study treatment. Participants will be asked to bring back the used empty antibiotic packs.

Blood to be sent for white cell count and C-reactive protein

Chest X-ray

c- Unscheduled Visits - Besides the two planned visits, participants will be allowed to contact the study team between the time points if they develop any of the symptoms of recurrence mentioned above. A study clinician will determine whether a clinical review is required and will arrange accordingly

#### Outcomes

# Primary outcome:

Incidence of failure of treatment as judged by trial clinician requiring further antibiotics and/or tube drainage and/or surgical intervention by six weeks post initial admission. Failure will be determined based on the one or more of the following parameter: clinical (recurrence of symptoms), biochemical (worsening of WCC [by 2000/mm $^3$ ] or CRP [by  $\geq$  20%] from discharge values) and radiological (chest X-ray +/- TUS evidence of increasing or new pleural collection).

# Secondary outcomes:

- Total length of antibiotic treatment (in days) in the study arms
- Number of participants with worsening in the 6-week chest X-ray as compared to discharge chest X-ray in the study arms. Chest X-ray pairs (discharge vs 6-week) will be read by a respiratory physician blinded to treatment allocation who will judge whether there is worsening (versus stability or improvement)
- Time (in days) to return to normal daily activities in participants of the study arms

Readmission within 30 days from discharge

# Sample Size:

This is a feasibility study and therefore no formal power calculation has been made. A sample size of 50 participants (25 per arm) was chosen by the study team simulating sizes chosen by trials examining outcomes in pleural infection in adult<sup>[8]</sup> and paediatric<sup>[13]</sup> populations.

### Randomisation and treatment allocation

Patients will be randomised 1:1 to the active or the control arm. The permuted block randomisation method will be used and the sequence will be generated using the online platform Sealedenvelop.com. At the point of randomisation, a member of the study team will log into the website and obtain the treatment allocation after confirmation of eligibility criteria. Being an open label study, allocation will be known to the patient and the study team performing assessments of study visits.

# Data management

Data will be collected directly into paper case report forms that will bear the study number of the participants but no other identifiable information. No data sources (e.g. lab results, etc.) will be stored within the trial files to maintain confidentiality of patients' medical data.

A screening log will be kept electronically on a spreadsheet that is password protected on a secure computer. This log will have the name and demographics of patients approached for the study as well as study number and treatment allocation for randomised patients.

At completion of study assessments for the last recruited patients, data will be transferred from paper CRFs to electronic form (spreadsheets) to allow statistical analysis. These spreadsheets will be stored securely after trial conclusion with the principal investigator and will be accessible to other members of the study team. Request to access study data by other teams will be expected via email and access will be granted by the principal investigator if the request is deemed reasonable.

#### **Statistics**

A per protocol analysis will be carried out for all outcomes. Given that this is a feasibility study, no replacement for participants lost to follow up will be attempted. Continuous variables will be compared between the study arms using t-test or Mann Whitney test according to the normality of the study data. Categorical variables (including primary outcome measure) will be compared using the Chi squared test or Fisher exact test as appropriate.

# Safety monitoring reporting

The study intervention (shorter antibiotic course) is envisaged to cause less adverse events due to less exposure to antibiotics. All treatment-related adverse events will be collected

routinely as part of the study. As a safety measure, an interim analysis will be planned when half the recruitment target is reached to ensure that the study intervention does not impose unacceptable risks to subjects randomised to this arm.

#### **Ethics and dissemination**

Approval will be sought from the Ethics Committee of Alexandria Faculty of Medicine and the protocol will be registered in an open-access trials database before the recruitment of the first patient. All participants will be required to sign an informed consent form prior to enrolment in the study. A scientific report with the results of the study will be prepared once the recruitment finishes.

#### References

- 1. Davies HE, Davies RJO, Davies CWH, on behalf of the BTS Pleural Disease Guideline Group. Management of pleural infection in adults: British Thoracic Society pleural disease guideline 2010. Thorax 2010;65(Suppl 2):ii41–53.
- 2. Cargill TN, Hassan M, Corcoran JP, Harriss E, Asciak R, Mercer RM, et al. A systematic review of comorbidities and outcomes of adult patients with pleural infection. Eur Respir J 2019;
- 3. Maskell NA, Lee YCG, Gleeson FV, Hedley EL, Pengelly G, Davies RJO. Randomized trials describing lung inflammation after pleurodesis with talc of varying particle size. Am J Respir Crit Care Med 2004;170(4):377–82.
- 4. Corcoran JP, Psallidas I, Gerry S, Piccolo F, Koegelenberg CF, Saba T, et al. Prospective validation of the RAPID clinical risk prediction score in adult patients with pleural infection: the PILOT study. Eur Respir J 2020;
- 5. Bedawi EO, Hassan M, Rahman NM. Recent developments in the management of pleural infection: a comprehensive review. The Clinical Respiratory Journal 2018;12(8):2309–20.
- 6. Hassan M, Cargill T, Harriss E, Asciak R, Mercer RM, Bedawi EO, et al. The microbiology of pleural infection in adults: a systematic review. European Respiratory Journal 2019;54(3):1900542.
- 7. Bhatnagar R, Maskell N. The modern diagnosis and management of pleural effusions. BMJ 2015;h4520.
- 8. Hooper CE, Edey AJ, Wallis A, Clive AO, Morley A, White P, et al. Pleural irrigation trial (PIT): a randomised controlled trial of pleural irrigation with normal saline versus standard care in patients with pleural infection. Eur Respir J 2015;46(2):456–63.
- 9. Porcel JM, Ferreiro L, Rumi L, Espino-Paisán E, Civit C, Pardina M, et al. Two vs. three weeks of treatment with amoxicillin-clavulanate for stabilized community-acquired complicated parapneumonic effusions. A preliminary non-inferiority, double-blind, randomized, controlled trial. Pleura and Peritoneum [Internet] 2020 [cited 2020 Sep 6];5(1). Available from: https://www.degruyter.com/view/journals/pp/5/1/article-20190027.xml
- 10. Rahman NM, Kahan BC, Miller RF, Gleeson FV, Nunn AJ, Maskell NA. A Clinical Score (RAPID) to Identify Those at Risk for Poor Outcome at Presentation in Patients With Pleural Infection. Chest 2014;145(4):848–55.
- 11. Chan A-W, Tetzlaff JM, Altman DG, Laupacis A, Gøtzsche PC, Krleža-Jerić K, et al. SPIRIT 2013 Statement: Defining Standard Protocol Items for Clinical Trials. Ann Intern Med 2013;158(3):200.
- 12. Kim SY, Flory J, Relton C. Ethics and practice of Trials within Cohorts: An emerging pragmatic trial design. Clinical Trials 2018;15(1):9–16.
- 13. Tagarro A, Otheo E, Baquero-Artigao F, Navarro M-L, Velasco R, Ruiz M, et al. Dexamethasone for Parapneumonic Pleural Effusion: A Randomized, Double-Blind, Clinical Trial. J Pediatr 2017;185:117-123.e6.